CLINICAL TRIAL: NCT01886898
Title: Growth of Infants Fed Starter Formula Containing Oligo-saccharides and the Probiotics Bifidobacterium & Lactobacillus
Brief Title: Synbiotics and Growth
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 05.23.INF
Record Dates: First submitted 2013-06-24; First posted 2013-06-26 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2013-06

CONDITIONS: Infants Growth
MeSH Terms: interventions — Infant Formula; Lactation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Standard starter infant formula (Placebo Comparator): starter infant formula from enrollment till 16 weeks of age
  Interventions: Other: Infant formula
- starter infant formula with prebiotics (Experimental): starter infant formula from enrollment till 16 weeks of age
  Interventions: Other: Infant formula
- starter infant formula with pro and prebiotics (Experimental): starter infant formula from enrollment till 16 weeks of age
  Interventions: Other: Infant formula
- breastfeeding group (Other): exclusively breastfeeding during the first 16 weeks of age
  Interventions: Other: Breastfeeding

INTERVENTIONS:
Other: Infant formula — infant formula
  Arms: Standard starter infant formula; starter infant formula with prebiotics; starter infant formula with pro and prebiotics
Other: Breastfeeding
  Arms: breastfeeding group

SUMMARY:
The primary objective of the trial is to assess the growth of the infants enrolled into the study. Other parameters to be measured include microbiota balance and certain blood biochemical values. In addition the infants' digestive tolerance of the formulae and frequency of morbidity will be investigated.

DETAILED DESCRIPTION:
The infants will be recruited between birth and 14 days of life and will start on the allocated study formula as soon as they are enrolled. In practice this will tend to be immediately after birth. The treatment period, in terms of data necessary for the primary outcome, will be until they reach 16 weeks old. Growth and other measurements will be collected on five separate occasions during this period, ie 2, 4, 8, 12 and 16 weeks of life. Although the study intervention formally ends at 16 weeks, it will be useful to have a follow up visit at 26 weeks to collect further data on the gut microflora in the sub-group of infants who have already provided a stool sample at 8 weeks. This follow-up visit will be of benefit to the subject as they receive a weight check and clinical examination by a paediatrician and will be offered to all subjects (no invasive procedures will be carried out).

ELIGIBILITY:
Inclusion Criteria:

* Healthy new-born infant
* Infant is less14 days old on day of enrollment
* Birthweight between 2500g and 4500g
* Gestational age over 37 weeks
* Singleton birth
* Infant's mother, before the 14th day of the child's life, has elected not to breastfeed
* Infant randomized in to a treatment group can expected to be exclusively fed the formula from enrolment until 16 weeks old
* Having obtained his/her legal representative's informed consent

Exclusion Criteria:

* Currently participating in another clinical trial
* Congenital illness or malformation that may affect normal growth
* Significant pre-natal and/or post-natal disease
* Re-hospitalisation for more than 2 days in the first 14 days of life. (Exceptionally, infants re-hospitalized because of jaundice may be enrolled in the study).
* Receiving antibiotic treatment at time of enrolment or in the 5 previous days.
* Receiving infant formula containing probiotics and/or prebiotics at the time of enrolment

Max Age: 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 311 (Actual)
Dates: Start 2007-06; Primary Completion 2009-02 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
mean weight gain (g/day) | over 16 weeks

SECONDARY OUTCOMES:
length (cm), head circumference (cm) | over 1 year
• digestive tolerance (stool characteristics and frequency, vomiting, spitting up, frequency of colic) | over 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto di Ostetricia e Genecologia, Palermo, Italy

REFERENCES:
- [Derived] Meli F, Puccio G, Cajozzo C, Ricottone GL, Pecquet S, Sprenger N, Steenhout P. Growth and safety evaluation of infant formulae containing oligosaccharides derived from bovine milk: a randomized, double-blind, noninferiority trial. BMC Pediatr. 2014 Dec 20;14:306. doi: 10.1186/s12887-014-0306-3. PMID 25527244